CLINICAL TRIAL: NCT01284244
Title: A Randomized Controlled Trial of the Uresta Continence Pessary; Short-term Uresta Efficacy Study (SURE Study)
Brief Title: A Randomized Controlled Trial of the Uresta Continence Pessary
Acronym: SURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Danny Lovatsis, Dr., Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100131A
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence, Stress; pessary; conservative management
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uresta (Experimental)
  Interventions: Device: Uresta pessary
- Silastic vaginal ring (Sham Comparator)
  Interventions: Device: Silastic ring

INTERVENTIONS:
Device: Uresta pessary — Participants randomized to the Uresta group will be fitted with device before immediately before performing the pad test. The Uresta pessary is made of medical grade rubber that has been extensively tested for safety. It is bell-shaped, with a narrow tip that allows for easy insertion into the vagina in a similar fashion to a tampon. The device can be easily inserted, and removed by a patient for use when needed. The Uresta comes in 3 sizes. Fitting starts with insertion of the smallest size. If urine leakage continues with valsalva or a cough stress test, it can be replaced by one size larger, until leakage is stopped. If the device prevents the patient from being able to void or is uncomfortable due to its size, the smaller size is replaced. Following the pad test, the participant will be given the opportunity to keep the device for continued use, or remove it if desired.
  Arms: Uresta
Device: Silastic ring — The silastic ring is a plastic flexible ring similar to that used to administer vaginal estrogen (Estring). It is well tolerated and would not contain any medications. Immediately before performing the pad test, it would be placed high in the vagina, away from the urethra. It would be removed immediately after the pad test. Draping will conceal from the patient which device was inserted.
  Arms: Silastic vaginal ring

SUMMARY:
Stress urinary incontinence (SUI) is defined as the involuntary loss of urine with an increase in abdominal pressure, caused either by a loss of support under the bladder neck, or intrinsic urethral sphincter deficiency. It is a common problem in women that can significantly impact quality of life, with up to 30% developing SUI at some point in their lifetime.

The most commonly utilized treatments for SUI include either pelvic floor (Kegel) exercises, or surgery. Many women find Kegel exercises unsatisfactory, but are reluctant to undergo a surgical procedure. Also, women who are poor candidates for surgery have limited options if Kegel exercises are unsuccessful. Over the years, there have been numerous attempts to develop effective non-surgical alternatives for treating SUI, but the results have been variable and the available data on efficacy limited.

A new intravaginal incontinence pessary (Uresta) has been developed for treating stress incontinence, and is currently available in Canada via a medical distributor. The self-positioning device is initially fitted by a healthcare provider, but then can subsequently placed by the patient as needed. Uresta is designed to be easily inserted into the vagina and spontaneously fall into position, providing support beneath the urethra. A single, uncontrolled study of 21 women showed that Uresta significantly reduces urinary incontinence measures, with no reported complications. Using questionnaires, a 47% reduction in self-reported SUI symptoms was demonstrated. Pad weight following a pad test, an objective assessment of urine loss, showed a 50% reduction in leakage.

This trial is intended to be a short-term assessment of the efficacy of the Uresta device, using a placebo arm in order to remove any of the possible sources of patient biases. The placebo ("sham") group will be obtained by placing a flexible silastic ring (inactivated Estring) high in the vagina where it will not alter urethral forces. The aim is to unequivocally determine whether the Uresta device provides the necessary urethral support to stop urine leakage from stress incontinence.

The hypothesis is that the Uresta device will significantly reduce urinary losses from baseline, shown as a significant reduction pad weight following a pad test with the device in place.

ELIGIBILITY:
Inclusion Criteria:

* Urodynamic diagnosis of stress urinary incontinence

Exclusion Criteria:

* Urodynamic diagnosis of mixed incontinence
* Bladder capacity less than 300mls
* Post-void residual over 100mls
* Pelvic organ prolapse greater than POP-Q stage 2
* Hematuria
* Undiagnosed vaginal bleeding
* Current pregnancy
* Previous incontinence or prolapse surgery
* Failed use of an incontinence pessary
* Physically unable to perform the activities included in the pad test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Lovatsis, MD MSc, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Department of Obstetrics and Gynecology, Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Farrell SA, Baydock S, Amir B, Fanning C. Effectiveness of a new self-positioning pessary for the management of urinary incontinence in women. Am J Obstet Gynecol. 2007 May;196(5):474.e1-8. doi: 10.1016/j.ajog.2006.11.038. PMID 17466709

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uresta | Silastic Vaginal Ring
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uresta | Silastic Vaginal Ring | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 50 (7) | 51 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: A 50% Reduction in Pad Test Weight
Description: A pad test is an objective measure of urine loss. With a full bladder, while wearing a pad, the participant completes five repetitions of the following physical activities: coughing, step climbing, heel bounce, standing from a sitting position and walking 50 yards. The weight of the pad is then determined.
  The primary outcome variable will be the achievement of a 50% reduction in the pad weight before and after device placement. This figure is obtained from the study by Farrell et al, where pad weight decreased from 20 grams to 9 grams with the use of the Uresta device.
Time Frame: Immediately after device placement (short term).
Measure: Count of Participants; unit: Participants
Arm/Group | Uresta | Silastic Vaginal Ring
Number analyzed (Participants) | 18 | 18
Participants | 12 | 4

ADVERSE EVENTS:
Arm/Group | Uresta | Silastic Vaginal Ring
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No